CLINICAL TRIAL: NCT03718260
Title: PSMA-PET Registry for Recurrent Prostate Cancer
Acronym: PREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Cancer Care Ontario (Other); Centre for Probe Development and Commercialization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4826
Record Dates: First submitted 2018-10-17; First posted 2018-10-24 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Prostate Cancer
Keywords: Prostate Cancer; Biochemical Failure; Node positive; PSMA-PET; [18F]DCFPyL PET/CT imaging; Radical Prostatectomy; Radiation Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Men who are node positive or who have persistently detectable PSA after initial radical prostatectomy will be restaged with [18F]-DCFPyL PET/ CT scan (PSMA PET)
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)
- Cohort 2 (Experimental): Men with biochemical failure after initial prostatectomy will be restaged with [18F]-DCFPyL PET/ CT scan (PSMA PET)
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)
- Cohort 3 (Experimental): Men with biochemical failure after initial radical prostatectomy and salvage radiotherapy will be restaged with [18F]-DCFPyL PET/ CT scan (PSMA PET)
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)
- Cohort 4 (Experimental): Men with biochemical failure after initial radical prostatectomy with or without adjuvant/ salvage radiotherapy who are currently on salvage hormone therapy will be restaged with [18F]-DCFPyL PET/ CT scan (PSMA PET)
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)
- Cohort 5 (Experimental): Men who have prior PSMA directed treatment for oligometastatic disease, such as lesion directed therapy (e.g. stereotactic radiosurgery) or systemic therapy (e.g. hormone therapy or chemotherapy) with subsequent biochemical failure will be restaged with [18F]-DCFPyL PET/ CT scan (PSMA PET)
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)
- Cohort 6 (Experimental): Men with biochemical failure after primary radiation therapy (external beam, brachytherapy or combinations together with or without hormone therapy) will be restaged with [18F]-DCFPyL PET/ CT scan (PSMA PET)
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)
- Cohort 7 (Experimental): [18F]-DCFPyL as a problem-solving tool in patients with prostate cancer when confirmation of the site of disease and/or disease extent may impact clinical management. Patients in this cohort require approval from an independent adjudication by Cancer Care Ontario.
  Interventions: Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET)

INTERVENTIONS:
Diagnostic Test: [18F]-DCFPyL PET/ CT scan (PSMA PET) — Participants will undergo re-staging with [18F]-DCFPyL PET/CT Scan (PSMA PET).

SUMMARY:
This study aims to institute a province-wide registry leveraging the availability of a new Positron Emission Tomography tracer, [18F]-DCFPyL and PET expertise across Ontario centers to improve our ability to characterize patterns of recurrence and personalize therapies in men with recurrent prostate cancer after primary treatment.

DETAILED DESCRIPTION:
This registry study will provide Ontario centres access to a new Positron Emission Tomography (PET) tracer, [18F]-DCFPyL, to improve our ability to identify areas of prostate cancer recurrence in men who have undergone surgical removal of their prostate gland (radical prostatectomy) or radiation of their prostate (external beam radiation, brachytherapy or a combination of both) and there is a suspicion of recurrence of the cancer. Men with suspected persistent or recurrent disease can be identified on the basis of a rising Prostate Specific Antigen (PSA) blood test, or the presence of node positive disease at the time of their surgery, or a PSA blood test continues to be detectable within 3 months after their surgery. It is the aim of this study to determine if [18F]-DCFPyL PET/CT can potentially identify areas of prostate cancer recurrence not seen with usual imaging (bone scan/CT scans) and impact the management of the disease. A report of the results of the [18F]-DCFPyL PET/CT will be provided to the participating physicians to determine a treatment plan. As part of the patient eligibility for [18F]-DCFPyL PET/CT participating physicians will complete a questionnaire after the [18F]-DCFPyL PET/CT information is provided to report how the results impact patient management. Actual interventions following completion of the [18F]-DCFPyL PET/CT will be tracked by linkage to provincial registries. Six centres across Ontario will participate in the registry study which is expected to take 4 years to complete with an additional one year of follow-up to capture patient outcomes.

PREP Phase 2 was initiated to investigate the hypothesis that conventional imaging is not adding to the information provided by PSMA PET/CT alone. PREP Phase 2 will retain the same study design as Phase I but will remove bone scan and computed tomography as criteria for entry into the study except for those patients with higher PSA (>10 ng/ml).

Identical cohort sizes will be accrued in Phase 2 to permit comparison of detection rates with similar confidence intervals with and without conventional imaging. Transition to PREP Phase 2 occurred when overall accrual to PREP exceeded 80% of target.

ELIGIBILITY:
Phase 2

Inclusion Criteria:

1. Written informed consent obtained
2. Male, Age ≥ 18 years
3. Prior primary treatment for prostate cancer with curative intent such as radical prostatectomy or radiotherapy for localized prostate cancer. Unless PET/CT requested as part of Cohort 7.
4. Suspected persistent or recurrent disease defined as one of the following (unless PET/CT requested as part of Cohort 7):

   1. High risk disease at the time of radical prostatectomy characterized by pathologically involved node(s) or persistently detectable PSA (>0.1ng/ml) within 3 months post-surgery
   2. Primary treatment for prostate cancer and biochemical failure (BF) with current management according to the following:

   i. Following primary radical prostatectomy, BF is defined as rising PSA on at least 2 occasions measured at least 1 month apart and with the most recent PSA measured at >0.1 ng/ml

   ii. Following primary radiotherapy for localized disease, BF is defined according to the Phoenix Definition, which is rising PSA on at least 2 occasions measured at least 1 month apart and with the most recent PSA measured greater than the nadir PSA + 2.0 ng/ml
5. Patient scenario falls into one of the 7 pre-defined cohorts. When patient scenario falls outside cohorts 1-6 participation in the Registry must be approved through the established CCO adjudication process for Cohort 7.
6. Karnofsky performance status 70 or better (ECOG 0, 1).
7. If PSA >10 mg/mL, conventional imaging consisting of bone scan and abdo-pelvic CT scan within 3 months of registration that is either equivocal, negative (no lesions) or positive for oligometastatic disease (4 or fewer unequivocal lesions identified).

Exclusion Criteria:

1. Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components.
2. Prior PSMA PET scan within 6 months of enrollment.
3. Patient cannot lie still for at least 60 minutes or comply with imaging.
4. Patients falling outside of Cohorts 1-6 where independent adjudication by CCO does not support participation in the Registry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be male (prostate cancer)
Enrollment: 3070 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of disease detection on PSMA PET | 5 years
  Phase 1: The number of men with detectable lesions on PSMA PET who have suspected recurrent or persistent disease post radical prostatectomy with or without adjuvant or salvage pelvic radiotherapy or hormone therapy as well as men treated with primary radiotherapy will be measured
  Phase 2: The number of men with detectable lesions on PSMA PET who have suspected recurrent or persistent disease post radical prostatectomy with or without adjuvant or salvage pelvic radiotherapy or hormone therapy as well as men treated with primary radiotherapy will be measured when PSMA PET/CT is used without routine pre-screening with conventional imaging.

SECONDARY OUTCOMES:
To determine correlations between PSA levels at time of imaging and presence of disease detected on PSMA PET. | 5 years
  The likelihood of disease detected on PSMA PET will be correlated with absolute PSA level at the time of PSMA PET as supplied on the eligibility form.
Proportion of men with oligometastatic recurrence (four or fewer sites including the prostate bed if positive) confirmed on PSMA PET/CT | 5 years
  Number of men with four or fewer sites of disease detected on PSMA PET
Number of men who have their management plan changed because of PSMA PET results | 5 years
  The number of men who have a change in management as indicated by responses from referring physicians on an impact questionnaire completed after PSMA PET scans are reported.
To determine the actual management delivered within 6 months of PSMA PET | 5 years
  Actual management within 6 months will be determined through linkage to existing health information registries and will include:
  1. Delivery of radiotherapy (anatomic site, dose and fractionation) - Cancer Care Ontario
  2. Biopsy of suspected recurrences (anatomic site, histology) - Provincial pathology database
  3. Use of salvage lymph node dissections - CIHI
  4. Use of salvage hormonal therapy/androgen deprivation
Compare PSA response at 6 months against PSA at the time of PSMA PET | 5 years
  PSA response will be examined by comparing 6 month PSA against PSA at the time of PSMA PET through the Ontario Laboratory Information Services and correlated with actual management as determined in Outcome 5.
Compare the detection rates of PSMA PET/CT when conventional imaging is used as part of the eligibility criteria (PREP) versus when conventional imaging is omitted (PREP Phase 2) | 5 years
  Number of men with detectable lesions as determined in the primary objective for PREP will be compared to the number of men with detectable lesions as determined in primary objective for PREP Phase 2.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, FRCPC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Ur Metser, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (6):
- Canada (6):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Basso Dias A, Finelli A, Bauman G, Veit-Haibach P, Berlin A, Ortega C, Avery L, Metser U. Impact of 18F-DCFPyL PET on Staging and Treatment of Unfavorable Intermediate or High-Risk Prostate Cancer. Radiology. 2022 Sep;304(3):600-608. doi: 10.1148/radiol.211836. Epub 2022 May 24. PMID 35608445
- [Derived] Metser U, Zukotynski K, Mak V, Langer D, MacCrostie P, Finelli A, Kapoor A, Chin J, Lavallee L, Klotz LH, Hagerty M, Hildebrand C, Bauman G. Effect of 18F-DCFPyL PET/CT on the Management of Patients with Recurrent Prostate Cancer: Results of a Prospective Multicenter Registry Trial. Radiology. 2022 May;303(2):414-422. doi: 10.1148/radiol.211824. Epub 2022 Jan 25. PMID 35076300